CLINICAL TRIAL: NCT02978742
Title: Evaluating and Implementing a Smartphone Application Treatment Program for Bulimia Nervosa and Binge Eating Disorder
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not funded.
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Aaron Keshen, Psychiatrist, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 59093009
Record Dates: First submitted 2016-11-29; First posted 2016-12-01 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Eating Disorder; Bulimia Nervosa; Binge Eating Disorder
Keywords: Eating Disorders; Bulimia Nervosa; Binge Eating Disorder; App; Smartphone; Self-Help; Coaching; Recovery Record; Mobile Phone; Cognitive Behavioral Therapy
MeSH Terms: conditions — Feeding and Eating Disorders; Bulimia Nervosa; Binge-Eating Disorder; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coached Recovery Record App (Experimental): Participants will complete the 8-week adaptive Recovery Record app program and will be linked with a healthcare professional who will provide standardized coaching, in the way of feedback and support to participants for the duration of the program.
  Interventions: Behavioral: Adaptive Recovery Record App; Behavioral: Standardized Coaching
- Uncoached Recovery Record App (Active Comparator): Participants will complete the 8-week adaptive Recovery Record app program on their own (i.e., without a coach providing feedback and support).
  Interventions: Behavioral: Adaptive Recovery Record App

INTERVENTIONS:
Behavioral: Adaptive Recovery Record App — Participants will use the Recovery Record smartphone app, which is a meal monitoring tool, that incorporates discrete reminders, motivational tools, social support, summative feedback, and coping skill suggestions. Participants will also receive tailored, algorithm-generated content in a structured manner that mimics the progression of psychotherapy (e.g., checking in with users, reminding them of their reasons for wanting to recover, and working towards goals) over the course of 8 weeks.
Behavioral: Standardized Coaching — Coaches (dietitians or mental health clinicians) will review patients' logs daily and participants will receive one communication of standardized feedback each day through the app based on their food records. A standardized feedback manual to be used by coaches has been developed by co-investigators (two PhD psychologists and one psychiatrist), and all feedback will be monitored for consistency and quality by co-investigators.
  Arms: Coached Recovery Record App

SUMMARY:
Bulimia nervosa and binge eating disorder pose a public health concern due to their high co-occurrence with other psychiatric disorders and poor physical health outcomes. It is therefore concerning that less than half of these patients seek treatment for their condition. People may be reluctant to seek treatment due to not wanting to disclose symptoms to family members. Even for those who do wish to seek help, treatment is often inaccessible due to the geographic centralization of eating disorder specialists and a low ratio of specialists to patients. Therefore, the aim of this study is to test a potential solution to these problems and make eating disorder care more private and accessible.

One possible way to improve the accessibility of treatment is through smartphone applications (or "apps"). We are testing an app called Recovery Record, which is primarily a tool used to self-monitor eating habits, where patients record their meals and related thoughts, feelings, emotions, and behaviours (e.g., binge eating/purging). The app also offers additional features such as discrete reminders to log meals, positive reinforcement, social support, coping strategy suggestions, and linking users with clinicians for real-time feedback and suggestions. The application is scientifically supported and has been tested with positive results.

Recently, app developers have created a computer-automated 8-week treatment program that uses the patient's data to provide a tailored and individualized treatment program. This program aims to mimic the process of therapy by checking in with users, reminding them of their reasons for wanting to recover, and working towards goals. We will be testing this automated app treatment program, comparing it both with and without input from a trained coach providing individualized feedback to users.

DETAILED DESCRIPTION:
The prevalence of bulimia nervosa (BN) is approximately 1.0-1.5% among women. With consistently higher prevalence rates, binge eating disorder (BED) affects up to 3.5% of women and 1.5% of men. These eating disorders represent a public health concern due to the high comorbidity of BN and BED with other psychiatric disorders and the association with poor physical health outcomes.

Given this public health impact, it is concerning that less than half of BN and BED patients seek treatment for their eating disorder. This is especially concerning since a greater duration of untreated illness is associated with a poorer prognosis. Individuals' reluctance to seek treatment is likely due to factors such as an avoidance of disclosing symptoms to family members or clinicians. For example, one study reported that 27% of adolescents with BN declined participation because they did not want their families involved. Even for those who do wish to engage, treatment is often inaccessible due to the geographic centralization of eating disorder specialists and a low ratio of specialists to patients.

Given the ubiquity of smartphone devices among adults and adolescents, one possible way to improve treatment accessibility and privacy is to offer it through a smartphone app. In recent development, an evidence-based smartphone app called Recovery Record (RR) has been conceived for use by people suffering from eating disorders as an adjunct to clinical treatment. This tool allows patients to self-monitor eating behaviours, connect with their clinician directly through the app, and provides other therapeutic features (e.g. cues coping skill use). Preliminary findings suggest that the app is feasible, with 67% of users continuing to log meals at 30 days. As well, RR is currently the most downloaded, most rated, and highest rated app of its kind, which suggests it is highly acceptable among users.

In support of these findings, one study demonstrated that 26% of app users in a clinically severe range at baseline demonstrated clinically significant reductions in eating disorder symptoms at least 28 days later, which is consistent with other forms of self-help for BN. Moreover, 89% of users reported that using Recovery Record helped their condition from getting worse and a majority reported improvements to the frequency of disordered behaviours, reported urges, and mood.

App developers have outfitted the app with an adaptive 8-week program that automatically uses patient data to tailor treatment for individual users (i.e. an automated pure self-help course of treatment). Although pure self-help is efficacious for BN and BED, self-help augmented by coaching (from a health care profession) has been associated with even better outcomes (with a moderate effect size). Given the support for this smartphone app and this potential avenue for providing private and accessible care to Nova Scotians, the aim of this study is to assess the efficacy of this adaptive smartphone app program, both coached and uncoached, for BN and BED patients.

ELIGIBILITY:
Inclusion Criteria:

* DSM-V diagnosis of bulimia nervosa or binge eating disorder
* Ages 16-65 years
* Has an Apple or Android smartphone with a data plan or daily access to Wi-Fi
* Is able to download smartphone applications from the Apple App Store or Google Play Store to their smartphone
* Lives in Canada
* Provides consent to participate

Exclusion Criteria:

* Actively engaged in psychological treatment, specifically for bulimia nervosa or binge eating disorder
* Lacks English fluency
* High risk for suicide, as determined by the Columbia Suicide Severity Rating Scale (Self-Report Screening Version)

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Change in Eating Disorder Symptom Severity | Measured at start of treatment, end of treatment (up to 8 weeks), and 3-month follow-up
  Self-reported symptom severity will be assessed with the Eating Disorder Examination Questionnaire (EDE-Q).

SECONDARY OUTCOMES:
Change in Binge Eating and Purging Frequency | Measured at start of treatment, end of treatment (up to 8 weeks), and 3-month follow-up
  Binge/purge frequency for the month prior will be gathered from self-reported EDE-Q responses.
Change in Clinical Impairment | Measured at start of treatment, end of treatment (up to 8 weeks), and 3-month follow-up
  The Clinical Impairment Assessment (CIA) will be used to identify changes in psychosocial impairment related to the participant's eating disorder.
Treatment Satisfaction | Measured at end of treatment (up to 8 weeks)
  Likert-scale and open-ended questions specific to the intervention will be used to assess participant satisfaction with treatment.
Treatment Adherence | Measured from start of treatment to the end of treatment (up to 8 weeks)
  Treatment completion will be defined as completing more than 75% of the 8-week treatment program and treatment dropout will be defined as completing any less than 75% of the program.

OTHER OUTCOMES:
Diagnosis of Bulimia Nervosa or Binge Eating Disorder | Pre-Screening
  A DSM-V diagnosis of bulimia nervosa or binge eating disorder will be determined with the Eating Disorder Diagnostic Scale (EDDS).
Suicidality | Pre-Screening
  Risk of suicide will be determined with the Columbia - Suicide Severity Rating Scale, Self-Report Screening Version (C-SSRS).

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Keshen, MD, FRCPC, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Capital Health District Health Authority, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tregarthen JP, Lock J, Darcy AM. Development of a smartphone application for eating disorder self-monitoring. Int J Eat Disord. 2015 Nov;48(7):972-82. doi: 10.1002/eat.22386. Epub 2015 Jul 27. PMID 26213130
- See also: Recovery Record Smartphone Application Website — http://www.recoveryrecord.com